CLINICAL TRIAL: NCT00790673
Title: A Phase 1/2, Randomized, Double-blind, Placebo-controlled, Dose-escalation Study Evaluating the Safety, Tolerability, Biological Activity, and Pharmacokinetics of Orally Administered CF102 in Subjects With Chronic Hepatitis C Genotype 1
Brief Title: A Phase 1/2 Study of CF102 in Patients With Chronic Hepatitis C Genotype 1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Can-Fite BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CF102-103HCV
Record Dates: First submitted 2008-09-17; First posted 2008-11-13 (Estimated); Results first posted 2015-04-15 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C; Viral hepatitis
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — 2-chloro-N(6)-(3-iodobenzyl)adenosine-5'-N-methyluronamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): CF102 1 mg qd
  Interventions: Drug: CF 102
- 2 (Experimental): CF102 1 mg bid
  Interventions: Drug: CF 102
- 3 (Experimental): CF102 1 mg bid; 16 weeks
  Interventions: Drug: CF 102
- 5 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CF 102 — Oral capsules
  Other Names: Cl-IB-MECA
  Arms: 1; 2; 3
Drug: Placebo — Matching placebo capsules
  Arms: 5

SUMMARY:
This trial will test the hypothesis that CF102 can safely and effectively suppress viral load in patients with chronic hepatitis C and high circulating levels of virus. The trial will monitor the safety of twice-daily oral dosing with CF102 over a 16-week period; will measure changes in viral load during therapy; and will measure blood concentrations of CF102 at various time points during dosing.

DETAILED DESCRIPTION:
This is a Phase 1/2, randomized, double-blind, placebo-controlled, dose-escalation study of subjects with chronic hepatitis C genotype 1. Eligible subjects will be assigned in a 3:1 ratio (8 subjects in each cohort) to receive qd or bid treatment for 15 days with oral CF-102 or with placebo. Dose escalation will occur in 2 sequential cohorts.

The decision to continue dosing within a cohort (eg, Subcohort 1a to Subcohort 1b), or to escalate to a new dose level Cohort (eg, Subcohort 1b to Subcohort 2a) will be determined by a blinded independent review of safety data. This review will be conducted by a qualified Safety Review Committee comprising the medical monitor, the consulting toxicologist, and an independent expert clinician.

For the first 2 cohorts, subjects will return to the study center for follow-up assessments on Days 8, 15, and 22. Subjects dosed qd will receive a total of 15 doses of CF-102. Subjects dosed bid will receive a total of 29 doses. The 30th dose has been deleted to accommodate PK sampling on the morning of Day 16, 24 hours after the last dose of CF-102.

For the 3rd cohorts, subjects will return to the study center for follow-up assessments on weeks 2, 4, 8, 12, 16 and 18.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 60 years of age
2. Body mass index ≤ 30 kg/m2
3. Either:

   1. no evidence of cirrhosis, or liver fibrosis corresponding to Metavir Stages 0 to 31 on a liver biopsy performed within the past 2 years, or
   2. a score of F0 or F1 on ActiTest-FibroTest performed within the past year.
4. Child-Pugh score ≤ 5 at Screening
5. Serologic evidence of chronic hepatitis C-infection (anti-HCV in serum)
6. HCV plasma RNA ≥ 1 x 105 IU/mL on 2 separate samples obtained during the screening period.
7. HCV genotype 1
8. The following laboratory values must be documented within the Screening period:

   * Hemoglobin > 11.0 g/dL for females and > 12.0 g/dL for males
   * Platelet count > 50 x109/L
   * Normal serum creatinine
   * Aspartic aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5-fold the upper limit of normal
   * International normalized ratio (INR) ≤ 1.3-fold normal
   * Serum albumin ≥ 3.6 gm/dL
9. Female subjects cannot be pregnant or breastfeeding and must be either postmenopausal, surgically sterile, abstinent, or using 2 proven methods of birth control
10. Sexually active male subjects must be practicing acceptable methods of contraception (eg, vasectomy, use of condom plus spermicide, monogamous relationship with a female partner who practices an acceptable method of contraception) during the treatment period
11. Negative serum ß-human chorionic gonadotropin (HCG, females of child-bearing potential only)
12. Provide informed consent
13. Willing to comply with all study requirements

Exclusion Criteria:

1. Positive test at Screening for human immunodeficiency virus
2. Uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4), angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack, or pulmonary embolism within 3 months prior to initiation of study drug
3. History of or ongoing cardiac dysrhythmias requiring treatment, atrial fibrillation of any grade, or persistent prolongation of the corrected QT (QTc) (Fridericia) interval to > 450 msec for males or > 470 msec for females
4. Positive results for drugs of abuse at Screening
5. Donation or loss of more than 400 mL blood within 2 months prior to anticipated dose administration
6. Participation in a clinical study with an investigational drug, biologic, or device within 3 months prior to anticipated dose administration
7. Previous exposure to CF102(Cohorts 1 and 2 only)
8. Males whose female partner is pregnant
9. Serum alpha-feto-protein > 50 ng/mL at screening
10. Any severe, acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, may interfere with the informed consent process and/or with compliance with the requirements of the study, or may interfere with the interpretation of study results and, in the investigator's opinion, would make the patient inappropriate for entry into this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2009-07; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Silverman, MD, Study Director — Can-Fite BioPharma Ltd
Locations (1):
- Rabin Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Bar-Yehuda S, Stemmer SM, Madi L, Castel D, Ochaion A, Cohen S, Barer F, Zabutti A, Perez-Liz G, Del Valle L, Fishman P. The A3 adenosine receptor agonist CF102 induces apoptosis of hepatocellular carcinoma via de-regulation of the Wnt and NF-kappaB signal transduction pathways. Int J Oncol. 2008 Aug;33(2):287-95. PMID 18636149
- See also: Can-Fite BioPharma — http://www.canfite.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 CF102 1 mg qd: CF102 1 mg qd
  CF 102: Oral capsules
- Cohort 2 CF102 1 mg Bid: CF102 1 mg bid
  CF 102: Oral capsules
- Cohort 3 CF102 1 mg Bid: CF102 1 mg bid; 16 weeks
  CF 102: Oral capsules
Period: Overall Study
Arm/Group | Cohort 1 CF102 1 mg qd | Cohort 2 CF102 1 mg Bid | Cohort 3 CF102 1 mg Bid | Placebo
Started | 6 | 6 | 12 | 8
Completed | 6 | 6 | 12 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 CF102 1 mg qd | Cohort 2 CF102 1 mg Bid | Cohort 3 CF102 1 mg Bid | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 12 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (12.7) | 54.5 (8.43) | 48.3 (12.4) | 42.1 (11.2) | 47.3 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 7 | 3 | 16
  Male | 3 | 3 | 5 | 5 | 16

OUTCOME MEASURES:

1. Primary Outcome: Adverse Event Profile of Repeated Dosing of CF102
Time Frame: 16 weeks
Measure: Number; unit: participants
Arm/Group | Cohort 1 CF102 1 mg qd | Cohort 2 CF102 1 mg Bid | Cohort 3 CF102 1 mg Bid | Placebo
Number analyzed (Participants) | 6 | 6 | 12 | 8
participants | 6 | 2 | 2 | 4

2. Primary Outcome: Effect of Viral Load
Time Frame: 16 weeks
Reporting Status: Not Posted

3. Primary Outcome: Pharmacokinetic Behavior of CF102 During Repeated Dosing
Time Frame: 16 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Evaluation of the Relationship Between Biomarkers of Peripheral Blood Mononuclear Cell Adenosine 3 Receptor (A3R) Expression and Clinical Effects
Time Frame: 16 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Cohort 1 CF102 1 mg qd | Cohort 2 CF102 1 mg Bid | Cohort 3 CF102 1 mg Bid | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/12 | 0/8
Other Adverse Events (participants affected / at risk) | 6/6 | 2/6 | 2/12 | 4/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 CF102 1 mg qd (N=6) | Cohort 2 CF102 1 mg Bid (N=6) | Cohort 3 CF102 1 mg Bid (N=12) | Placebo (N=8)
Fatigue (General disorders) | 2 (6) | 0 (0) | 0 (0) | 0 (0) — Fatigue
HEADACHE (Nervous system disorders) | 4 (6) | 2 (6) | 2 (12) | 4 (8) — HEADACHE
Palpitations (Cardiac disorders) | 2 (6) | 0 (0) | 0 (0) | 0 (0) — Palpitations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No